CLINICAL TRIAL: NCT02163889
Title: Serial Therapeutic and Antifungal Monitoring Protocol
Acronym: STAMP
Status: Completed | Type: Observational
Sponsor: T2 Biosystems (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-00254
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2015-09

CONDITIONS: Candidemia
Keywords: Candida; Blood culture; Antifungal therapy; Sepsis
MeSH Terms: conditions — Candidemia; Torulopsis; Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — At each time point, three 4 ml whole blood specimens will be collected. One sample will be tested, and the remaining samples will be available for use in investigating discrepant T2Candida assay and blood culture results, or may be used for research purposes
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Candida Positive Patients: Symptomatic adult patients, confirmed via blood culture with species identification to be positive for Candida

SUMMARY:
The objective of this study is to investigate T2Candida performance as a monitoring tool for post-therapy clearance of Candida compared to blood culture.

This study will collect a T2clinical specimen and companion blood culture from patients who have exhibited a positive blood culture by gram stain for yeast, and who are receiving treatment with antifungal therapy.

DETAILED DESCRIPTION:
One blood culture and one set of T2clinical specimens will be collected at specified intervals to monitor the clearance of Candida infection from the bloodstream.

Each T2 result will be compared to the companion blood culture result. The comparison will determine if the presence of antifungal therapy inhibits blood culture and leads to an incidence of blood culture false negative test results. The T2 result, which is not impacted by the presence of antifungal therapy, can show that the pathogen is still present for some additional period of time.

ELIGIBILITY:
Inclusion Criteria:

* Subject or subject's authorized representative must be able to understand, read and sign the study specific informed consent form after the nature of the study has been fully explained to them.
* Subject is between 18-95 years of age
* Subject has a blood culture result that is positive for yeast within 36 hours of enrollment

Exclusion Criteria:

* Subject has other co-morbid condition(s) that, in the opinion of the Investigator, could limit the subject's ability to participate in the study or impact the scientific integrity of the study
* All T2 Bio individual clinical research specimens contain < 3 ml of blood
* Use of any novel (i.e. not commercially available) drug compound within 30 days prior to the collection of T2 Bio blood specimens.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving treatment with antifungal therapy for 1 of 5 Candida species:
  * Candida albicans
  * Candida tropicalis
  * Candida glabrata
  * Candida parapsolosis
  * Candida krusei
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Time to negative test result | 14 days post enrollment
  The number of days to a negative test result will be compared between the T2Candida Test and blood culture.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Alabama, Birmingham, Alabama
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island

REFERENCES:
- [Derived] Mylonakis E, Zacharioudakis IM, Clancy CJ, Nguyen MH, Pappas PG. Efficacy of T2 Magnetic Resonance Assay in Monitoring Candidemia after Initiation of Antifungal Therapy: the Serial Therapeutic and Antifungal Monitoring Protocol (STAMP) Trial. J Clin Microbiol. 2018 Mar 26;56(4):e01756-17. doi: 10.1128/JCM.01756-17. Print 2018 Apr. PMID 29367293